CLINICAL TRIAL: NCT07345871
Title: Investigating the Effectiveness of Connective Tissue Dry Needling Technique on Patients With Low Back Pain Caused by Local Pain at Superior Posterior Iliac Spine: a Single-blind, Randomized Controlled Trial
Brief Title: Connective Tissue Dry Needling for Low Back Pain Related to Local Posterior Superior Iliac Spine Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Mohammad Javaherian, Principal Investigator, University of Social Welfare and Rehabilitation Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USWR-3441
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain (CLBP); Sacroiliac Joint Dysfunction; Mechanical Low Back Pain
Keywords: Mechanical Low Back Pain; Sacroiliac Joint Dysfunction; Connective Tissue Disorders; Dry Needling; Fascia / Fascial Manipulation
MeSH Terms: conditions — Low Back Pain; Connective Tissue Diseases | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise therapy (Active Comparator): Participants in this group will receive only the standardized exercise program over two weeks.
  Interventions: Procedure: Exercise therapy
- CTDN (Mahshid technique) plus Exercise therapy (Experimental): Participants in this group will receive CTDN targeting the PSIS region together with the standardized exercise program over two weeks.
  Interventions: Procedure: Connective tissue dry needling; Procedure: Exercise therapy

INTERVENTIONS:
Procedure: Connective tissue dry needling — Connective tissue dry needling: Eight sterile single-use needles placed 1.5 cm from the PSIS center, inserted at about 45° to bony contact, withdrawn 0.5 cm, rotated five times to maximal tissue stiffness, then retained for 20 minutes with concurrent infrared therapy. Three sessions per week for two weeks, total six sessions. Needle size 50 mm × 0.5 mm.
  Arms: CTDN (Mahshid technique) plus Exercise therapy
Procedure: Exercise therapy — Pelvic bridging, leg-lowering, curl-up or bridging, and isolated lumbar stabilizer training. Three sets of ten repetitions for each exercise, three sessions per week for two weeks.

SUMMARY:
This single-blind randomized controlled trial will aim to determine the effectiveness of a connective tissue dry needling (CTDN) technique, in reducing pain and improving function in individuals with chronic mechanical low back pain associated with pain and tenderness at the posterior superior iliac spine (PSIS). Forty participants with local PSIS-related low back pain will be recruited and randomly assigned into two groups using the block balanced randomization method. The treatment group will receive CTDN targeting connective tissue trigger points around the PSIS in addition to a sacroiliac joint stabilization exercise program, while the control group will perform the same exercise program alone under the supervision of a physiotherapist. The intervention protocol will span two weeks, during which participants will attend three treatment sessions per week, for a total of six sessions. The primary outcome measurement will use the Visual Analog Scale (VAS) to assess pain intensity. The study will measure secondary outcomes through lumbar range of motion (ROM) in flexion and extension and pressure pain threshold (PPT), and Roland-Morris Disability Questionnaire (RMDQ) functional disability and Short Form-36 (SF-36) health-related quality of life. The researchers will assess all outcomes at three time points: baseline and after the first session, and the sixth session, while VAS will receive an additional assessment at the 3-month follow-up. The findings of this study are expected to provide evidence supporting CTDN as a safe, effective, and cost-efficient treatment option for PSIS-related mechanical low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most widespread musculoskeletal disorders, which creates substantial disability and healthcare expenses throughout both developed and developing nations (1,2). The medical field categorizes LBP into two distinct types: specific and non-specific. The medical field identifies specific LBP through detectable causes, including infections and trauma and structural problems but non-specific LBP lacks identifiable spinal pathology and represents most cases (3,4). Research shows that LBP originates from multiple sources including intervertebral discs and facet joints and sacroiliac joints (SIJ) and their associated ligaments and muscles (5-8).

Research indicates that the SIJ acts as a primary pain source for 15-25% of patients who experience chronic LBP (9). The SIJ plays a vital biomechanical role by connecting the spine to the lower extremities through its complex network of ligaments and fascia which distributes both axial and rotational forces (10). The Posterior Superior Iliac Spine (PSIS) represents a significant anatomical reference point near the SIJ where multiple essential soft tissue structures including the long posterior sacroiliac ligament and thoracolumbar fascia and gluteus maximus converge (10,11). Studies based on clinical and anatomical evidence show that tissue dysfunction or irritation in this area leads to pain development in the PSIS region (12).

The Fascial Distortion Model (FDM) among other recent models demonstrates how fascia-bone junctions produce musculoskeletal pain through their mechanical interactions. The model indicates that extended periods of inactivity together with abnormal mechanical forces disrupt cellular communication and mineral transport at these junctions which leads to fascial adhesions and persistent pain (13,14). The complex anatomy and high sensitivity of the PSIS area has led to increased research about treatments that focus on the surrounding connective tissue structures.

The minimally invasive technique of dry needling fascial structures known as fascia dry needling (FDN) aims to create mechanical and cellular changes in the extracellular matrix of connective tissues. Research shows that dry needling procedures in connective tissue areas lead to increased fibroblast activity and cytoskeletal rearrangement which may create better matrix organization and decrease pain signals (15,17-19). Research through imaging and mechanobiological studies has proven that needle rotation in both directions leads to substantial tissue movement and increased gene expression for tissue repair without inflicting any structural harm (20-25).

Research conducted with animal subjects has validated these mechanistic results through observations of tendon recovery and tissue reorganization following needling procedures (22-25). The clinical application of dry needling has produced beneficial results for patients with lateral epicondylosis and Achilles tendinopathy and thoracic pain syndromes by improving their pain levels and mobility and functional abilities (26,29,30).

The medical field lacks any randomized controlled trial that investigates how fascia dry needling affects the PSIS region despite rising evidence about dry needling effects on different musculoskeletal conditions. The current clinical guidelines recommend periarticular or intra-articular injections for PSIS or SIJ-related pain but these procedures come with high costs and complex procedures and potential adverse effects for patients (31). The non-invasive nature of FDN makes it an attractive treatment option which needs thorough clinical assessment.

The research study aims to evaluate PSIS area fascia dry needling as an additional treatment for standard physiotherapy represents a critical knowledge gap in current medical literature. The confirmation of safety and effectiveness of this treatment method would lead to updated clinical guidelines and help decrease reliance on invasive procedures while giving healthcare providers an effective new treatment option for patients with PSIS-related mechanical low back pain.

Hypotheses:

Null Hypothesis (H₀): The fascia dry needling technique (Mahshid method) has no significant effect on pain intensity, lumbar range of motion, pain pressure threshold, functional disability, or quality of life in patients with chronic mechanical low back pain and point tenderness at the posterior superior iliac spine.

Alternative Hypothesis (H₁): The fascia dry needling technique (Mahshid method) has a significant positive effect on pain intensity, lumbar range of motion, pain pressure threshold, functional disability, and quality of life in patients with chronic mechanical low back pain and point tenderness at the posterior superior iliac spine.

ELIGIBILITY:
Inclusion criteria:

1. Adults aged 18 to 75 years.
2. Diagnosed with chronic mechanical low back pain localized at the posterior superior iliac spine region.
3. Presence of point tenderness reproducible by palpation at the posterior superior iliac spine area.
4. Pain duration of at least two weeks, indicating the non-acute stage of low back pain.
5. Negative results in at least three out of five sacroiliac pain provocation tests (Distraction, Compression, Thigh Thrust, Sacral Thrust, Gaenslen).
6. Pain intensity ≥ 3 on the Numeric Rating Scale at baseline.
7. Ability to communicate and cooperate with the research team during intervention and follow-up.
8. Access to WhatsApp or equivalent communication application for follow-up pain reporting at the 3-month stage.

Non-inclusion criteria:

1. Presence of lumbar radicular pain or referred pain to the lower limbs.
2. History of lumbar spine trauma within the previous three months.
3. Fear or intolerance of needling procedures.
4. Current use of anticoagulant medication.
5. Known lymphatic disorders, immunosuppressive diseases, or neurological conditions such as epilepsy or seizure disorders.
6. Pregnancy or suspected pregnancy.

Exclusion criteria:

1. Voluntary withdrawal of consent at any time during the study.
2. Inability to tolerate the intervention or adverse reaction during treatment sessions.
3. Occurrence of serious adverse events or complications (e.g., infection, bleeding).
4. Non-compliance with treatment protocol or missing more than two sessions.
5. Any intercurrent illness or therapy that could interfere with the study outcomes or safety assessment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-04-10 (Estimated); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest value, representing the most severe pain.
Visual Analog Scale | 30 minutes
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest value, representing the most severe pain.
Visual Analog Scale | 2 weeks
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest value, representing the most severe pain.
Visual Analog Scale | 3-month follow-up
  It is a commonly used tool for measuring pain. The patient is asked to mark their pain level on a 100-mm line, and the marked distance is then measured with a ruler from the left end and recorded. The scale typically ranges from zero, indicating no pain, to the highest value, representing the most severe pain.

SECONDARY OUTCOMES:
Lumbar flexion range of motion | Baseline
  Lumbar flexion will be measured using a digital inclinometer app (iHandy® Level, version 1.70.3, Apple Inc.) installed on an iPhone® 8 Plus device. The device will be placed on the L1 and S2 spinous processes while the participant performs maximal flexion. The total range of motion will be calculated by subtracting the S2 angle from the L1 angle.
Lumbar flexion range of motion | 30 minutes
  Lumbar flexion will be measured using a digital inclinometer app (iHandy® Level, version 1.70.3, Apple Inc.) installed on an iPhone® 8 Plus device. The device will be placed on the L1 and S2 spinous processes while the participant performs maximal flexion. The total range of motion will be calculated by subtracting the S2 angle from the L1 angle.
Lumbar flexion range of motion | 2 weeks
  Lumbar flexion will be measured using a digital inclinometer app (iHandy® Level, version 1.70.3, Apple Inc.) installed on an iPhone® 8 Plus device. The device will be placed on the L1 and S2 spinous processes while the participant performs maximal flexion. The total range of motion will be calculated by subtracting the S2 angle from the L1 angle.
Lumbar extension range of motion | Baseline
  Lumbar extension will be measured using a digital inclinometer app (iHandy® Level, version 1.70.3, Apple Inc.) installed on an iPhone® 8 Plus device. The device will be placed on the L1 and S2 spinous processes while the participant performs maximal extension. The total range of motion will be calculated by subtracting the S2 angle from the L1 angle.
Lumbar extension range of motion | 30 minutes
  Lumbar extension will be measured using a digital inclinometer app (iHandy® Level, version 1.70.3, Apple Inc.) installed on an iPhone® 8 Plus device. The device will be placed on the L1 and S2 spinous processes while the participant performs maximal extension. The total range of motion will be calculated by subtracting the S2 angle from the L1 angle.
Lumbar extension range of motion | 2 weeks
  Lumbar extension will be measured using a digital inclinometer app (iHandy® Level, version 1.70.3, Apple Inc.) installed on an iPhone® 8 Plus device. The device will be placed on the L1 and S2 spinous processes while the participant performs maximal extension. The total range of motion will be calculated by subtracting the S2 angle from the L1 angle.
Pressure Pain Threshold at the posterior superior iliac spine Region | Baseline
  Pressure Pain Threshold will be measured using a mechanical pressure algometer (Lutron FG-5020, Taiwan). Pressure will be applied vertically over the posterior superior iliac spine region at a rate of approximately 1 kg/s until the participant first reports pain. The value will be recorded in kg/cm². Higher scores indicate greater tolerance and lower tissue tenderness.
Pressure Pain Threshold at the posterior superior iliac spine Region | 30 minutes
  Pressure Pain Threshold will be measured using a mechanical pressure algometer (Lutron FG-5020, Taiwan). Pressure will be applied vertically over the posterior superior iliac spine region at a rate of approximately 1 kg/s until the participant first reports pain. The value will be recorded in kg/cm². Higher scores indicate greater tolerance and lower tissue tenderness.
Pressure Pain Threshold at the posterior superior iliac spine Region | 2 weeks
  Pressure Pain Threshold will be measured using a mechanical pressure algometer (Lutron FG-5020, Taiwan). Pressure will be applied vertically over the posterior superior iliac spine region at a rate of approximately 1 kg/s until the participant first reports pain. The value will be recorded in kg/cm². Higher scores indicate greater tolerance and lower tissue tenderness.
Roland-Morris Disability Questionnaire | Baseline
  The Roland-Morris Disability Questionnaire is a 24-item validated self-reported questionnaire assessing the impact of low back pain on daily life. Each "Yes" response scores 1 point, while "No" scores 0, yielding a total between 0 and 24. Higher scores indicate greater disability.
Roland-Morris Disability Questionnaire | 30 minutes
  The Roland-Morris Disability Questionnaire is a 24-item validated self-reported questionnaire assessing the impact of low back pain on daily life. Each "Yes" response scores 1 point, while "No" scores 0, yielding a total between 0 and 24. Higher scores indicate greater disability.
Roland-Morris Disability Questionnaire | 2 weeks
  The Roland-Morris Disability Questionnaire is a 24-item validated self-reported questionnaire assessing the impact of low back pain on daily life. Each "Yes" response scores 1 point, while "No" scores 0, yielding a total between 0 and 24. Higher scores indicate greater disability.
Short Form-36 Health Survey | Baseline
  The validated Persian version of SF-36 will be used to assess eight domains of health-related quality of life (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health). Scores range from 0 (worst) to 100 (best).
Short Form-36 Health Survey | 30 minutes
  The validated Persian version of SF-36 will be used to assess eight domains of health-related quality of life (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health). Scores range from 0 (worst) to 100 (best).
Short Form-36 Health Survey | 2 weeks
  The validated Persian version of SF-36 will be used to assess eight domains of health-related quality of life (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health). Scores range from 0 (worst) to 100 (best).

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided yet, but at this moment, we have decided to share brief data with future researchers after requesting and submitting ethical committee permission.

REFERENCES:
- [Result] Langevin HM, Churchill DL, Fox JR, Badger GJ, Garra BS, Krag MH. Biomechanical response to acupuncture needling in humans. J Appl Physiol (1985). 2001 Dec;91(6):2471-8. doi: 10.1152/jappl.2001.91.6.2471. PMID 11717207
- [Result] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Result] Vlaeyen JWS, Maher CG, Wiech K, Van Zundert J, Meloto CB, Diatchenko L, Battie MC, Goossens M, Koes B, Linton SJ. Low back pain. Nat Rev Dis Primers. 2018 Dec 13;4(1):52. doi: 10.1038/s41572-018-0052-1. PMID 30546064
- [Result] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Result] Manchikanti L, Singh V, Pampati V, Damron KS, Beyer CD, Barnhill RC. Is there correlation of facet joint pain in lumbar and cervical spine? An evaluation of prevalence in combined chronic low back and neck pain. Pain Physician. 2002 Oct;5(4):365-71. PMID 16886014
- [Result] Yang H, Liu H, Li Z, Zhang K, Wang J, Wang H, Zheng Z. Low back pain associated with lumbar disc herniation: role of moderately degenerative disc and annulus fibrous tears. Int J Clin Exp Med. 2015 Feb 15;8(2):1634-44. eCollection 2015. PMID 25932092
- [Result] Vaccaro AR, Ring D, Scuderi G, Cohen DS, Garfin SR. Predictors of outcome in patients with chronic back pain and low-grade spondylolisthesis. Spine (Phila Pa 1976). 1997 Sep 1;22(17):2030-4; discussion 2035. doi: 10.1097/00007632-199709010-00018. PMID 9306535
- [Result] Werner CM, Hoch A, Gautier L, Konig MA, Simmen HP, Osterhoff G. Distraction test of the posterior superior iliac spine (PSIS) in the diagnosis of sacroiliac joint arthropathy. BMC Surg. 2013 Oct 31;13:52. doi: 10.1186/1471-2482-13-52. PMID 24175954
- [Result] Cohen SP. Sacroiliac joint pain: a comprehensive review of anatomy, diagnosis, and treatment. Anesth Analg. 2005 Nov;101(5):1440-1453. doi: 10.1213/01.ANE.0000180831.60169.EA. PMID 16244008
- [Result] Kiapour A, Joukar A, Elgafy H, Erbulut DU, Agarwal AK, Goel VK. Biomechanics of the Sacroiliac Joint: Anatomy, Function, Biomechanics, Sexual Dimorphism, and Causes of Pain. Int J Spine Surg. 2020 Feb 10;14(Suppl 1):3-13. doi: 10.14444/6077. eCollection 2020 Feb. PMID 32123652
- [Result] Barker PJ, Hapuarachchi KS, Ross JA, Sambaiew E, Ranger TA, Briggs CA. Anatomy and biomechanics of gluteus maximus and the thoracolumbar fascia at the sacroiliac joint. Clin Anat. 2014 Mar;27(2):234-40. doi: 10.1002/ca.22233. Epub 2013 Aug 20. PMID 23959791
- [Result] Murakami E, Kurosawa D, Aizawa T. Treatment strategy for sacroiliac joint-related pain at or around the posterior superior iliac spine. Clin Neurol Neurosurg. 2018 Feb;165:43-46. doi: 10.1016/j.clineuro.2017.12.017. Epub 2017 Dec 21. PMID 29306764
- [Result] Langevin HM, Churchill DL, Wu J, Badger GJ, Yandow JA, Fox JR, Krag MH. Evidence of connective tissue involvement in acupuncture. FASEB J. 2002 Jun;16(8):872-4. doi: 10.1096/fj.01-0925fje. Epub 2002 Apr 10. PMID 11967233
- [Result] Langevin HM, Bouffard NA, Badger GJ, Churchill DL, Howe AK. Subcutaneous tissue fibroblast cytoskeletal remodeling induced by acupuncture: evidence for a mechanotransduction-based mechanism. J Cell Physiol. 2006 Jun;207(3):767-74. doi: 10.1002/jcp.20623. PMID 16511830
- [Result] Langevin HM, Yandow JA. Relationship of acupuncture points and meridians to connective tissue planes. Anat Rec. 2002 Dec 15;269(6):257-65. doi: 10.1002/ar.10185. PMID 12467083